CLINICAL TRIAL: NCT03224416
Title: Effects of Acute Alcohol on Sex-Specific Delay Discounting and Subsequent Sexual Decision Making Among MSM
Brief Title: Individual and Contextual Factors That Influence Sexual Decisions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Mark Celio, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Project Now (Phase II)
Record Dates: First submitted 2017-03-13; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Binge Drinking; Unsafe Sex; HIV/AIDS; Sexually Transmitted Diseases
Keywords: Alcohol; Delay Discounting; Risky Sexual Behavior; Decision Making; MSM
MeSH Terms: conditions — Binge Drinking; Unsafe Sex; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Ethanol; Organization and Administration

STUDY DESIGN:
Intervention Model Description: The alcohol/placebo/nonalcohol design involves three conditions. In the alcohol condition (target BrAC = 0.080g%), the participant will be told he is receiving alcohol and will receive beverages of 1:4 parts vodka and tonic water with dashes of lime juice and mint, all mixed in his presence. In the placebo condition (target BrAC = 0.000g%), the participant will be told he is receiving alcohol but will receive beverages of 1:4 parts flat tonic water (served from a vodka bottle) and tonic water, with a minimal amount of vodka "floated" on the surface (using a lime juice bottle) to provide the smell and taste of vodka, with lime juice and mint, all mixed in his presence and served in glasses with vodka-soaked rims. In the true control (or nonalcohol) condition, the participant will be told he is receiving no alcohol and will be given water (poured in his presence) in a volume comparable to the other conditions.
Who Masked: Participant
Masking Description: Masking only applies to those participants who are randomly assigned to the placebo condition, which is described in detail above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alcohol (Experimental): In the alcohol condition (target BrAC = 0.080g%), the participant will be told he is receiving alcohol and will receive beverages of 1:4 parts vodka and tonic water with dashes of lime juice and mint, all mixed in his presence.
  Interventions: Other: Alcohol Administration
- Placebo (Placebo Comparator): In the placebo condition (target BrAC = 0.000g%), the participant will be told he is receiving alcohol but will receive beverages of 1:4 parts flat tonic water (served from a vodka bottle) and tonic water, with a minimal amount of vodka "floated" on the surface (using a lime juice bottle) to provide the smell and taste of vodka, with lime juice and mint, all mixed in his presence and served in glasses with vodka-soaked rims.
  Interventions: Other: Placebo Alcohol Administration
- True Control (Sham Comparator): In the true control (or nonalcohol) condition, the participant will be told he is receiving no alcohol and will be given water (poured in his presence) in a volume comparable to the other conditions.
  Interventions: Other: No Alcohol Administration

INTERVENTIONS:
Other: Alcohol Administration — In the alcohol condition (target BrAC = 0.080g%), the participant will be told he is receiving alcohol and will receive beverages of 1:4 parts vodka and tonic water with dashes of lime juice and mint, all mixed in his presence.
  Arms: Alcohol
Other: Placebo Alcohol Administration — In the placebo condition (target BrAC = 0.000g%), the participant will be told he is receiving alcohol but will receive beverages of 1:4 parts flat tonic water (served from a vodka bottle) and tonic water, with a minimal amount of vodka "floated" on the surface (using a lime juice bottle) to provide the smell and taste of vodka, with lime juice and mint, all mixed in his presence and served in glasses with vodka-soaked rims.
  Arms: Placebo
Other: No Alcohol Administration — In the true control (or nonalcohol) condition, the participant will be told he is receiving no alcohol and will be given water (poured in his presence) in a volume comparable to the other conditions.
  Arms: True Control

SUMMARY:
For decades, men who have sex with men (MSM) have carried the heaviest burden associated with the HIV epidemic in the United States. Although MSM represent a minority (i.e., approximately 4%) of the male population in the United States, in 2010 MSM accounted for 78% of new HIV infections among males. Furthermore, the estimated number of new HIV infections attributed to male-to-male sexual contact is currently rising. In order to improve interventions to decrease transmission of HIV among MSM, it is important to have a better understanding of predictors of risky sexual behavior. Alcohol use is among the most reliable predictors of risky sexual behavior. Unfortunately, studies of alcohol use and risky sex among MSM have mainly relied on survey-based methods that cannot advance our understanding of the causal mechanisms linking acute alcohol use to HIV risk behavior.

This study will utilize an "alcohol/placebo/nonalcohol" design to examine the mechanisms underlying the association between the acute effects of alcohol (i.e., pharmacological and expectancy) and risky sexual decision making in MSM. Focal mechanisms include sex-specific delay discounting (SSDD), and the core constructs of the Cognitive Mediation Model. The alcohol/placebo/nonalcohol design involves three conditions. In the alcohol condition (target BrAC = 0.080g%), the participant will be told he is receiving alcohol and will receive beverages of 1:4 parts vodka and tonic water with dashes of lime juice and mint, all mixed in his presence. In the placebo condition (target BrAC = 0.000g%), the participant will be told he is receiving alcohol but will receive beverages of 1:4 parts flat tonic water (served from a vodka bottle) and tonic water, with a minimal amount of vodka "floated" on the surface (using a lime juice bottle) to provide the smell and taste of vodka, with lime juice and mint, all mixed in his presence and served in glasses with vodka-soaked rims. In the true control (or nonalcohol) condition, the participant will be told he is receiving no alcohol and will be given water (poured in his presence) in a volume comparable to the other conditions. This 3-group design will enable us to test the pharmacological effects of alcohol while accounting for potential expectancy effects. Participants (Target N = 150-180) will be randomly assigned to one condition; all will undergo the same protocol, which will be completed within one experimental session. The study protocol consists of baseline assessment, followed by beverage administration, followed by post-drinking assessment of SSDD and sexual decision making, followed by debriefing.

DETAILED DESCRIPTION:
Significance and Specific Aims of Project

Men who have sex with men (MSM) continue to be disproportionately affected by the HIV epidemic in the United States. However, the experimental research designed to advance our knowledge of the causal link between alcohol use and risky sex has disproportionately focused on heterosexual men and women. Experimental studies are needed to test established theories and explore new mechanisms linking alcohol to HIV risk among MSM. This proposed project will experimentally test if sex-specific delay discounting (SSDD) is a mechanism of action underlying the association between alcohol and risky sexual behavior among MSM. More specifically stated, the aims are to:

1. Examine the pharmacological effect of alcohol on sex-specific delay discounting in MSM, with the prediction that individuals who consume alcohol will display greater sexual impulsivity
2. Examine the expectancy effect of alcohol on sex-specific delay discounting in MSM, with the prediction that those who receive placebo will evince greater sexual impulsivity than true controls
3. Test whether sex-specific delay discounting mediates the effects of alcohol on risky sexual decision making in MSM, using the CMM as a theoretical base for hypothesis testing

Participant Population

The participant population will consist of males age 21 to 35 years who are able to read and communicate in English. Eligible participants are: 1) single (i.e., not in a mutually monogamous relationship for at least 3 months); 2) sexually active as defined by any anal sex (i.e., receptive or insertive) with another man in the past 12 months; and 3) have had condomless anal sex with a male partner in their lifetime; 4) have had at least one sexual encounter with a male partner met online in their lifetime; 5) characterized as a current heavy drinker, as defined by self-report of one or more episodes of heavy drinking (i.e., ≥5 standard drinks in a single occasion) during the past 30 days; and 5) HIV negative, based on self-report.

Non-drinkers, light to moderate drinkers, and individuals with current alcohol problems (as indexed by an AUDIT score ≥16) or drug problems (as indexed by a DAST score ≥6) will be excluded. Given that this is a study of MSM, females will be excluded. Furthermore, individuals who do not meet the relationship status and sexual activity criteria above will be excluded. Lastly, individuals who participated in Phase 1 of this research program will be excluded from Phase 2 Based on recruitment rates from studies at Brown, the investigators estimate that one quarter of participants completing the screening consent will be eligible for the study. As such, the investigators plan to obtain screening consent from approximately 600 to 800 individuals with the hope of yielding 150 to 180 participants eligible for the experimental session.

Recruitment and Screening

Participants will be recruited using established and approved methods that have been applied in our community, including online advertisement through the Brown CAAS and Brown Alcohol Research Center on HIV (ARCH) websites, flyers posted at CAAS- and ARCH-affiliated clinical and community centers, and flyers posted at public venues and organizations in the local community. In addition to these direct recruitment strategies, this study will employ chain referral sampling (i.e., "snowball sampling"), in which project staff will ask men who respond to our advertisements if they would be willing to inform others about our study.

Project staff will also contact individuals who have completed the online survey for our research participant pool. The participant pool survey provides an efficient means to identify individuals who are interested in participating in research studies on sexual minority men's health. The HRPP confirmed that the procedures necessary for creating and managing this participant pool do not constitute human subjects research, and therefore do not require IRB review. The participant pool survey includes items that are sufficient to determine whether an individual meets preliminary screening criteria for the current study. As with our other recruitment strategies, all individuals recruited through the participant pool will be asked to complete the dedicated screening consent and survey to determine full eligibility for this study.

Methodology and Procedures

Screening. Upon contact, potential participants will be given a brief description of the study and will receive a link to our online screening consent form and screening survey. Upon completion of the screening survey, those who do not meet the inclusion criteria will be notified of their ineligibility online. Eligible participants will be contacted by a research assistant to describe the experimental session further and confirm their interest in participating. Eligible participants will be informed that the experimental session will last 2.5 hours, plus the time it takes for BrAC to fall to .02%. Participants will be told not to drive to the session; public transportation or cab vouchers will be provided if necessary. Participants will be asked to bring photo identification to their session, to avoid using alcohol or drugs that are not prescribed (including over-the-counter drugs) for 24 hours prior to their appointments, and to fast for 3 hours before their appointments. Participants agreeing to these terms will be scheduled for the experimental session.

Informed Consent Procedure. All experimental sessions will be conducted at CAAS in Providence, RI. Our labs are designed to facilitate studies involving alcohol administration. When participants arrive to the lab, the research assistant will review photo identification to verify the participant's age, then they will collect a BrAC to ensure that they are .000%. Those with a BrAC above .000% will be rescheduled. Next, the research assistant will review all sections of the informed consent document with the participant. The research assistant will ask the participant if he understands the key component involved in participation, and will answer any remaining questions before obtaining the participant's signature on the appropriate documentation. After obtaining consent, the research assistant will review a standard medical condition agreement, which asks participants to indicate whether they have any medical conditions or are taking any medications for which alcohol use is contraindicated. RAs will emphasize that questions are being asked of participants to ensure their safety, and inquire about whether there are any safety reasons why they should not participate. Lists of affected conditions and medications will be provided.

Experimental Session Protocol. Participants will be randomly assigned to one of three potential conditions described above. The research assistant will collect measures of the participant's weight and height for determining the volume of beverage to be administered. This includes determining the appropriate dose of alcohol for those assigned to the alcohol condition. Dose amounts will be calculated using a well-validated algorithm. Next participants will be asked to complete a baseline assessment battery via computer-delivered self-report questionnaire. Finally, the research assistant will encourage the participant to use the restroom prior to initiating experimental procedures.

After completing the baseline measures, participants will undergo the beverage administration protocol, which will be identical for all participants so as to avoid bias due to potential timing effects. Duration and timing of beverage administration and post-drinking assessment is based on pharmacokinetic assumptions that peak blood alcohol is approximately 60 minutes after consumption. Participants in the alcohol condition will consume a volume of alcohol to reach a peak BrAC of .080g%. The total volume will be divided into three drinks to be consumed over the course of 15 minutes. Following consumption, BrAC will be measured every 5-minutes, and post-drinking assessment will be initiated when the participant's BrAC is .035g%, as this corresponds with the initiation of stimulant effects of alcohol. The estimated absorption period to reach this level is 10 to 20 minutes. Initiation of post-drink assessment for placebo and true control participants will be determined using a yoked control design, such that each control participant is assigned to undergo the same waiting period and the same number of breath tests as a corresponding alcohol participant.

Upon reaching a BrAC of .035g% (or comparable time for placebo and control), participants begin the post-drinking assessment protocol, comprising an arousal prime, two measures of sex-specific delay discounting, followed by the MSM stimulus story. The instructions for each of these tasks will be computer-delivered, and participant responses will be collected via computer-based self-report questionnaires. Within the MSM scenario, participants are asked in open-ended format to respond to other character in the story or to describe what happens next. These responses will be audio recorded using a digital recording device set to automatically record when the participant begins speaking. Throughout this protocol, which will last approximately 35-45 minutes, BrAC will be measured every 10-15 minutes for all participants independent of condition. To evaluate the success of the experimental manipulation, subjective intoxication (e.g., "how intoxicated do you feel?") will be measured every 10-15 minutes as well.

Following the assessment phase, participants in the placebo and control conditions will be debriefed and provided with a taxi home. Participants in the alcohol condition will begin the recovery period, in which they will be able to eat a snack, use the restroom, and wait comfortably. BrAC will be assessed every 15-20 minutes until it is verified at .02g% or below, at which point they will be debriefed and provided with a taxi or public transportation home.

ELIGIBILITY:
Inclusion Criteria:

* single (i.e., not in a mutually monogamous relationship for at least 3 months)
* sexually active as defined by any anal sex (i.e., receptive or insertive) with another man in the past 12 months
* have had condomless anal sex with a male partner in their lifetime
* have had at least one sexual encounter with a male partner met online in their lifetime
* characterized as a current heavy drinker, as defined by self-report of one or more episodes of heavy drinking (i.e., ≥5 standard drinks in a single occasion) during the past 30 days; and 5) HIV negative, based on self-report.

Exclusion Criteria:

* Non-drinkers and light to moderate drinkers
* Individuals with current alcohol problems (as indexed by an AUDIT score ≥16)
* Individuals with current drug problems (as indexed by a DAST score ≥6)
* Females (as this is a study of men who have sex with men).

Ages: 21 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender males
Enrollment: 120 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Sexual Partner Delay Discounting Task | Approximately 20-30 minutes after beverage administration within our single-session, lab-based protocol.
  This delay discounting task measures hypothetical choice preference for immediately available sexual partners versus delayed but more attractive sexual partners. Data collected across 35 items is used to calculate a discounting rate, with a higher rate suggesting a more impulsive preference for immediate sexual activity.
Sex Discounting Task | Approximately 20-30 minutes after beverage administration within our single-session, lab-based protocol.
  This discounting task measures the degree to which the value of hypothetical condom-protected sex decreases as a product of the amount of time one would have to wait for a condom to be available. Data collected across 32 items is used to calculate a discounting rate, with a higher rate suggesting a more impulsive preference for immediate and condomless sexual activity.
Condomless Anal Sex Intentions | Approximately 45-50 minutes after beverage administration within our single-session, lab-based protocol.
  In the context of this laboratory-based experiment, participants read a hypothetical scenario depicting a sexual interaction with a casual sexual partner. Intention to have condomless anal sex with this partner is assessed in the middle and at the end of this scenario. Intention is rates as "yes" or "no" in response to the question "In this situation, do you have anal sex with [this partner] without a condom?"

SECONDARY OUTCOMES:
Perceived Sex Potential | Approximately 35 minutes after beverage administration within our single-session, lab-based protocol.
  In the context of this laboratory-based experiment, participants read a hypothetical scenario depicting a sexual interaction with a casual sexual partner. Perceives sex potential is assessed at the beginning of the scenario by asking "In this scenario, how likely are you to have sex tonight?" Participants respond using an 11-point scale with "0" anchored at "not at all likely" and "10" anchored at "very likely."
Perceived Sexual Risks and Benefits Scale | Approximately 40 minutes after beverage administration within our single-session, lab-based protocol.
  In the context of this laboratory-based experiment, participants read a hypothetical scenario depicting a sexual interaction with a casual sexual partner. Within the scenario, participants are asked "When thinking about whether or not to have sex with this partner tonight, would you consider each of the following reasons? Please mark YES if you would consider the reason, and NO if you would not consider it in this situation." The list comprises 34 items, including 17 perceived risks and 17 perceived benefits. For each risk and benefit endorsed, participants also rate the extent to which the reason would influence their decision using a 5-point scale, with "0" anchored at "not influential and "5" anchored at "extremely influential."
Online Sexual Communication | Approximately 45 minutes after beverage administration within our single-session, lab-based protocol.
  In the context of this laboratory-based experiment, participants read a hypothetical scenario depicting a sexual interaction with a casual sexual partner. During the scenario, the participant is asked "At this point in the story, would you want to talk about anything else before agreeing to meet?" Participants who answer"yes" are then asked "What else you would want to talk about? Please use the text boxes below to describe what else you want to talk about." Responses are open ended. Finally, participants are asked "Each of the topics you want to discuss with this partner are listed below. For each, please write down exactly how you would ask this partner on Grindr. If you would use emoji in your message, please describe which ones?" Again, responses are open ended. These data are qualitative in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Celio, PhD, Principal Investigator — 1979
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No